CLINICAL TRIAL: NCT00018746
Title: Efficacy of Threshold vs. Subthreshold TMS in the Treatment of Depression
Brief Title: Transcranial Magnetic Stimulation in Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MHBS-037-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation

SUMMARY:
The study examines efficacy of repetitive transcranial magnetic stimulation in treating severely depressed patients who are medicated.

DETAILED DESCRIPTION:
Medicated, treatment resistant, depressed patients are randomized to active or sham repetitive transcranial magnetic stimulation (rTMS). Responding patients go into a six months follow-up period.

ELIGIBILITY:
severe treatment-resistant depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hoffman; Dan Oren
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

REFERENCES:
- [Derived] Wu NQ, Gao Z, Zheng Y, Li W, Li JN, Xu HY, Cheng XS, Wu Y, Wang Y, Wang ZJ, Yang JG, Yang YJ; China Acute Myocardial Infarction Registry Study Group. [Status of intra-aortic balloon pump application and related factors in Chinese patients with acute myocardial infarction]. Zhonghua Xin Xue Guan Bing Za Zhi. 2018 Jan 24;46(1):26-31. doi: 10.3760/cma.j.issn.0253-3758.2018.01.005. Chinese. PMID 29374934
- [Derived] Fu R, Yang YJ, Dou KF, Yang JG, Gao XJ, Xu HY, Wu Y, Li W, Wang Y, Jia YL, Jin C; China Acute Myocardial Infarction Registry. [Age-related differences in the clinical symptoms and triggering factors among Chinese patients with acute myocardial infarction]. Zhonghua Xin Xue Guan Bing Za Zhi. 2016 Apr 24;44(4):298-302. doi: 10.3760/cma.j.issn.0253-3758.2016.04.005. Chinese. PMID 27112606